CLINICAL TRIAL: NCT06721000
Title: Patient Control Epidural Versus Conventional Epidural After Total Hip Replacement
Brief Title: Patient Control Epidural Versus Conventional Epidural.
Status: Enrolling by invitation | Type: Observational
Sponsor: Liaquat National Hospital & Medical College (Other)
Responsible Party: Principal Investigator, Uruba Shamshad, Dr Uruba, Liaquat National Hospital & Medical College
Other Study IDs: App # 0881- 2023- LNH - ERC
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Post Operative Pain, Acute; Sedation Score; Degree of Motor Block; Length of Hospital Stay; Amount of Analgesic Used
Keywords: Patient control epidural analgesia; Conventional epidural
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PCEA group: Epidural catheter is inserted and patient is given a remote to control the amount of drug given through patient control epidural pump.
- Non-PCEA group: Epidural catheter is inserted and the amount of drug set will be delivered via infusion pump.

SUMMARY:
As one of the complications of THR is post operative pain, which usually requires epidural catheter insertion.

We are comparing the effect of patient control epidural versus conventional epidural for patient's satisfaction.

DETAILED DESCRIPTION:
More than 20 years of successful usage of epidural analgesia for post operative pain treatment include intermittent provider-administer bolus, patient control analgesia and continuous epidural infusion with or without patient control epidural analgesia. The main drawback of conventional epidural infusion is that it does not allow for individual variation in management of pain. As a result, patient control epidural analgesia has replaced it in recent years.3. It has been demonstrated that continuous epidural infusion with patient control epidural analgesia is highly effective at providing consistent analgesia, improving patient satisfaction, and reducing the workload of anesthesia provider but it is linked to higher local anesthetic consumption4 In patient undergoing THR, patient control epidural analgesia may be considered as an appropriate alternative for managing post operative pain.

ELIGIBILITY:
Inclusion Criteria:

Age >18 years. ASA 1-2 on pre anesthesia evaluation. Spontaneous breathing. Spo2 >95% Informed consent for participation.

Exclusion Criteria:

A history of long-term opioid therapy (use of opioid analgesic at doses higher than codeine 120mg/day, hydrocodone 40mg/day, tramadol 200mg/day or oxycodone 40mg/day 0-4 days before surgery).

Indication of revision surgery during immediate post operative care. Acute skin disease. Patients' refusal. ASA 3 and 4. Hypersensitivity to study drugs.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient population will be from liaquat national hospital.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2025-01-25 (Estimated)

PRIMARY OUTCOMES:
Visual analogue score | 24 hours
  Patient satisfaction will be assessed after 2hours, 12hours and 24hours after surgery according to patient's pain intensity.
  Score will be from 1-10, 10 means maximum satisfaction and 1 means minimal satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Liaquat national hospital and medical college, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Considering patient's status of understanding i will decide it later.

REFERENCES:
- See also: Related Info — https://doi.org/10.5507/bp.2018.068